CLINICAL TRIAL: NCT07193758
Title: Return to Work After Lumbar Surgery for Radicular Pain: a Nationwide Survey of Spinal Surgeons' Practices and Perceptions
Brief Title: Return to Work After Lumbar Surgery: a Nationwide Survey of Spinal Surgeons' Practices
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70903
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Radicular Pain; Lumbar Surgery; Radicular Pain Related to Lumbosacral Disc Disease; Fusion of Spine, Lumbar Region; Disc Herniation With Radiculopathy; Lumbar Decompression
Keywords: Radicular pain; Lumbar surgery; Lumbar decompression; Lumbar discectomy; Lumbar fusion; Survey; Spinal surgeons; Return to work; Sick leave advice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Belgian spinal surgeons: Belgian spinal surgeons who are members of the Spine Society of Belgium (SSBe). The survey will be distributed through the SSBe membership list.

SUMMARY:
This national cross-sectional survey investigates the current practices and perceptions of Belgian spinal surgeons regarding return to work (RTW) after lumbar surgery for radicular pain. The study aims to (1) assess surgeons' advice on RTW and sick leave, (2) identify barriers and facilitators encountered when providing RTW guidance, and (3) explore how these factors relate to surgeon characteristics such as demographics, hospital setting, and professional experience. The results will inform clinical practice recommendations and support the development of targeted interventions to improve RTW guidance.

DETAILED DESCRIPTION:
Return to work (RTW) after lumbar surgery is shaped by a combination of medical, psychosocial, and system-level factors. Although clinical guidelines increasingly recognize RTW as an essential outcome, limited evidence exists on how surgeons address this issue in everyday practice and what challenges they encounter.

This national cross-sectional survey will be distributed to members of the Spine Society of Belgium (SSBe). It explores surgeons' demographics, current clinical practices regarding RTW advice and sick leave, communication strategies with patients, perceived professional roles and responsibilities, and barriers and facilitators in providing RTW guidance.

The findings will provide insights into current practices, highlight modifiable barriers, and support the development of evidence-based clinical recommendations and targeted interventions to optimize RTW guidance after lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgeons or neurosurgeons who perform lumbar surgery in Belgium.
* Members or affiliates of the Spine Society of Belgium (SSBe), as survey distribution will occur through the SSBe member list.
* Willing to participate in the survey, as evidenced by voluntary completion of the online questionnaire. Informed consent is implied after reading the participant information sheet.

Exclusion Criteria:

* Surgeons not performing lumbar surgery.
* Surgeons not affiliated with SSBe.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Belgian spinal surgeons (orthopaedic surgeons and neurosurgeons) who perform lumbar surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reported practices regarding return to work advice and sick leave following lumbar surgery | Through study completion, an average of 3 months (anticipated January 2026)
  Measured using a custom-designed online questionnaire. Topics include timing of advice, recommended duration of sick leave, and content of return-to-work guidance. Results reported as frequencies and percentages.

SECONDARY OUTCOMES:
Reported barriers and facilitators to providing return to work guidance | Through study completion, an average of 3 months (anticipated January 2026)
  Measured using multiple-choice and Likert-scale questions. Topics include professional-level barriers and facilitators. Results reported as frequencies, percentages, and mean Likert scores (1-5; higher = greater agreement).
Surgeon demographics and practice characteristics | Through study completion, an average of 3 months (anticipated January 2026)
  Demographic and professional background questions including age, sex, specialty, years in practice, hospital setting, and surgical case load. Results summarized as frequencies and percentages.
Reported confidence and perceived responsibility in discussing return to work | Through study completion, an average of 3 months (anticipated January 2026)
  Measured using 5-point Likert scale questions. Topics include self-reported confidence in discussing return-to-work and perceived responsibility among surgeons. Results reported as mean scores (1 = strongly disagree, 5 = strongly agree; higher scores = greater confidence/responsibility).

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Rummens, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
The study involves a small professional population (Belgian spinal surgeons), where sharing individual-level responses could risk indirect identification despite anonymization. Only aggregated, group-level results will be reported.